CLINICAL TRIAL: NCT03345498
Title: Study to Compare Virological Response to 0.5 mg Daily Versus 1.0 mg Daily Oral Doses of Entecavir in Chronic Hepatitis B Virus Infection Related Decompensated Cirrhosis
Brief Title: Entecavir for Decompensated HBV Cirrhosis
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-140-IMP-93
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis B; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis | interventions — entecavir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETV 0.5 mg: Group of study participants who were started on 0.5 mg/day of entecavir
  Interventions: Drug: Entecavir
- ETV 1.0 mg: Group of study participants who were started on 1.0 mg/day of entecavir
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Entecavir is the antiviral drug of choice recommended for hepatitis B virus treatment in presence of decompensated cirrhosis

SUMMARY:
Entecavir (ETV) and tenofovir (TDF) are the first-line drugs for treatment of chronic hepatitis B virus (HBV) infection. Chronic HBV infection gradually progress to liver cirrhosis. Over time, as liver damage and cirrhosis advance, the illness progress to a stage termed as decompensated cirrhosis, characterized by development of one or more of serious, life-threatening complications (ascites, hepatic encephalopathy, variceal bleeding or jaundice). In HBV related decompensated cirrhosis, antiviral treatment is shown to provide benefit.

For HBV related decompensated cirrhosis, EVT is the drug of choice as it has been shown to be effective and safe. The usual dose of ETV for chronic HBV infection is 0.5 mg orally once daily. Somehow, the recommended dose of ETV for decompensated cirrhosis has been 1.0 mg/d. The literature provides no justification for using this double dose of ETV. Since 0.5 mg daily works well in other stages of disease, there is little reason why it should not work well even in treatment-naïve decompensated cirrhosis. Considering the limitations of available literature, physicians' are divided in their opinion about the drug dose and are prescribing either of the two doses of ETV for this group. Hence, there is a need to assess whether the usual 0.5 mg/d of ETV would work as well as the 1.0 mg/d dose of ETV in decompensated cirrhosis due to HBV infection.

Investigators planned this open-labeled observational study with objective to compare the efficacy of HBV suppression achieved using 0.5 mg daily and 1.0 mg daily of ETV in HBV-related decompensated cirrhosis by comparing the mean reduction in HBV DNA level from baseline after 24 weeks of treatment.

In present study investigators propose to enroll 15 participants in each group who has been started on either doses (0.5 mg and 1.0 mg) of entecavir and measure serum HBV DNA levels in blood specimens (5 ml) will be collected at different time points, i.e. at baseline, 2, 4, 8, 12 and 24 weeks after starting entecavir.

DETAILED DESCRIPTION:
Background Chronic infection with hepatitis B virus (HBV), if untreated, may progress to liver cirrhosis, portal hypertension and hepatocellular carcinoma. Currently, oral administration of one of the nucleos(t)ide analogues (NAs) is the preferred treatment for chronic HBV infection. Of the five NAs approved for HBV treatment, lamivudine, adefovir and telbivudine are no longer preferred, and the recent guidelines from all three major international liver disease associations [American Association for the Study of Liver Disease (AASLD), European Association for Study of Liver (EASL), and Asia-Pacific Association for Study of Liver (APASL)] recommend the use of either entecavir (ETV) or tenofovir (TDF) as first-line drugs, because of their lower propensity to induce drug-resistant mutants and hence better efficacy.

Chronic liver disease due to any cause gradually progress to liver cirrhosis. Over time, liver damage and cirrhosis advances to a stage termed as decompensated cirrhosis, characterized by development of one or more of serious, life-threatening complications (ascites, hepatic encephalopathy, variceal bleeding or jaundice). Treatment of HBV infection with anti-viral drugs, in presence of decompensated cirrhosis, is beneficial.

In presence of HBV-related decompensated cirrhosis, EVT is the drug of choice as it has been shown to be effective and safe. The usual dose of ETV for chronic HBV infection is 0.5 mg orally once daily. Somehow, the recommended dose of ETV in presence of decompensated cirrhosis has been 1.0 mg/d. The literature provides little direct justification for using this double dose of ETV. Possibly, initially, ETV was used empirically in this dose to achieve a rapid HBV suppression in this high-risk group with prior exposure to lamivudine in advanced liver disease. However, since 0.5 mg daily works well in other stages of disease, there is little reason why it should not work well even in treatment-naïve decompensated cirrhosis. On the other hand, use of this higher dose of ETV adds to cost, a major consideration in areas where medical expenses are mostly met with out of the pocket expenses. Hene, in view of above-mentioned limitations of available literature, opinion of physicians is divided and either of the two doses of ETV is used in HBV related decompensated cirrhosis.

Hence, there is a need to assess whether the usual 0.5 mg/d of ETV would work as well as the 1.0 mg/d dose of ETV in decompensated cirrhosis due to HBV infection.

Hypothesis

Entecavir treatment in a dose of 0.5 mg once daily and of 1.0 mg daily have comparable antiviral efficacy in HBV-related decompensated cirrhosis.

Objective

To compare the efficacy of HBV suppression achieved using 0.5 mg daily and 1.0 mg daily of ETV in HBV-related decompensated cirrhosis by comparing the reduction in HBV DNA level from baseline till up to 24 weeks of treatment.

Study design

Open-label administration of 0.5 mg or 1.0 mg daily of entecavir for 24 weeks with comparison of mean reduction in HBV DNA levels from baseline in participants receiving the two dose schedules.

Study subjects

Participants with decompensated liver cirrhosis and replicative HBV infection (HBsAg positive, serum HBV DNA titer >100,000 IU/mL) will be enrolled, irrespective of their HBeAg and anti-HBe test results. Diagnosis of cirrhosis will be based on a combination of typical clinical, biochemical, radiological and endoscopic findings. Hepatic decompensation will be defined according to the most recent definition of APASL which defines it as significant liver dsyfunction as indicated by (i) raised serum bilirubin (more than 2.5 times the upper limit of normal) and prolonged prothrombin time (prolonged by more than 3 s or international normalized ratio >1.5) or (ii) occurrence of ascites or (iii) hepatic encephalopathy.

Participants with one or more of the following features will be excluded: (i) prior exposure to NAs or other specific treatment for HBV infection (e.g. pegylated interferon), (ii) hepatocellular carcinoma, (iii) co-infection with any other hepatotropic viruses or HIV, (iv) acute-on-chronic liver failure as defined by the criteria laid down by Asia-Pacific Association for the Study of Liver, (iv) significant alcohol intake or another concomitant hepatobiliary disease, (v) expected survival below 4 weeks (e.g. hemodynamic instability, active sepsis, hepatorenal syndrome, etc), (vi) use of immunosuppressive medication or (vii) portal vein thrombosis. Also, a participant who is not in a position to return for the scheduled follow-up visits will be excluded.

Study procedures

Enrollment and consent

We will consider to enroll the participants with HBV related decompensated cirrhosis and is planned for treatment, based on their clinical conditions, with either 0.5 or 1.0 mg daily doses of Entecavir by their treating physician. For those who agree to participate (by signing an informed consent), clinical and laboratory findings (including baseline HBV DNA level) will be recorded.

Follow-up and outcome measure

Blood specimens (5 ml) will be collected at different time points, i.e. at baseline, 2, 4, 8, 12 and 24 weeks after starting Entecavir. Serum will be separated and stored at -80C till analysis. In each specimen, HBV DNA will then be assessed using a quantitative real-time PCR.

Sample size

It is proposed to enroll 15 participants in each arm.

Data analysis

The rate of decline in HBV DNA levels with time will be compared between groups, using methods for longitudinal data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants with decompensated liver cirrhosis and
* Replicative HBV infection (HBsAg positive, serum HBV DNA titer >100,000 IU/mL) regardless of HBeAg and anti-HBe test results

Exclusion Criteria:

* prior exposure to NAs or other specific treatment for HBV infection (e.g. pegylated interferon)
* hepatocellular carcinoma
* co-infection with any other hepatotropic viruses or HIV
* acute-on-chronic liver failure as defined by Asia-Pacific Association for the Study of Liver criteria
* significant alcohol intake or another concomitant hepatobiliary disease
* expected survival below 4 weeks (e.g. hemodynamic instability, active sepsis, hepatorenal syndrome, etc)
* use of immunosuppressive medication or
* portal vein thrombosis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will consider to enroll the participants with HBV related decompensated CLD and is planned for treatment, based on their clinical conditions, with either 0.5 or 1.0 mg daily doses of Entecavir by the treating physician. For those who agree to participate (by signing an informed consent), clinical and laboratory findings (including baseline HBV DNA level) will be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percent reduction in quantitative HBV DNA levels at 2 weeks post-treatment | 2 weeks from start of ETV treatment
  Quantitative HBV DNA will be measured in study participants at 2 weeks post-treatment in participants receiving either intervention. Percent reduction at 2 weeks from baseline level will be compared between interventions.
Percent reduction in quantitative HBV DNA levels at 4 weeks post-treatment | 4 weeks from start of ETV treatment
  Quantitative HBV DNA will be measured in study participants at 2 weeks post-treatment in participants receiving either 0.5 mg or 1.0 mg daily doses of entecavir. HBV DNA will be measured after 2 weeks of ETV. Percent reductions at 4 weeks from baseline level will be compared.

SECONDARY OUTCOMES:
Percent reduction in quantitative HBV DNA levels at 8, 12 and 24 weeks post-treatment | 8, 12 and 24 weeks from start of ETV treatment
  Quantitative HBV DNA will be measured in study participants at 8,12 and 24 weeks post-treatment in participants receiving either intervention. Percent reduction at 8, 12 and 24 weeks from baseline level will be compared between interventions.
Change in disease severity as assessed by change in CTP score and change in MELD score | 24 weeks from start of ETV treatment
  Liver disease severity scores (Child-Turcotte-Pughscore and Model for End-stage Liver Disease (MELD) score will be assessed after 24 weeks of either intervention and change in score from baseline level will be compared between interventions

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goel, DM, Principal Investigator — Associate Professor, Gastroenterology
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goel A, Rungta S, Verma P, Verma A, Verma AN, Rai P, Aggarwal R. Viral suppression is comparable with 0.5 mg and 1.0 mg daily doses of entecavir in treatment-naive HBV-related decompensated cirrhosis. Antivir Ther. 2020;25(5):267-273. doi: 10.3851/IMP3375. PMID 33404519